CLINICAL TRIAL: NCT00164645
Title: Problem Solving for Caregivers of Patients With Traumatic Brain Injury
Brief Title: Problem Solving for Caregivers of Persons With Brain Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCIPC-00019101
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2005-09

CONDITIONS: Traumatic Brain Injury
Keywords: Emotional outcomes; health outcomes; traumatic brain injury; caregiving
MeSH Terms: conditions — Brain Injuries, Traumatic

INTERVENTIONS:
Behavioral: Problem Solving intervention

SUMMARY:
Family caregivers of persons with traumatic brain injury (TBI) have long-term demands that tax their coping abilities and adversely affect their health and well-being. This project will test the effectiveness of a problem-solving training program tailored to the unique needs of family caregivers of persons with TBI. Over a 3-year period, family caregivers and their care recipients will be recruited and randomly assigned to a problem-solving intervention group (n=40 dyads) or a control group (n=40 dyads). Participants in the problem-solving intervention group will receive four face-to-face problem-solving training sessions and monthly telephone problem-solving sessions over the course of 1 year. Control group participants will receive a handbook of educational materials and a staff member will contact each control group participant monthly by telephone to review these materials and other informational needs. No problem-solving training will be provided to control participants throughout the year.

Caregivers and care recipients will be assessed at four points during their participation: at the initial assessment, at 4 months, at 8 months, and at the completion of the 1-year participation period. All evaluations will be conducted in the participants' homes. Measures of problem-solving ability, caregiver burden, and adjustment (depression, health, satisfaction with life) will be collected. Structural equation modeling and other regression/inferential analyses will be used to determine the effects of problem solving on caregiver adjustment over time after taking into account care recipient adjustment and caregiver ethnicity. This project will: (1) demonstrate how specified physical and emotional outcomes of caregivers and care recipients are related to caregiver problem-solving abilities and how these relationships vary as a function of time; (2) evaluate the effectiveness of a community-based, problem-solving intervention that will be delivered to caregivers; and (3) identify caregivers and care recipients with TBI who are at risk for adverse emotional and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Minimum age of 19 years Brain injury diagnosis at least 6 mos in-house non-paid caregiver of person with brain injury functional literacy caregiver willing to discuss abuse issues

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Elliot, PhD, ABPP, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- See also: Related Info — http://www.uab.edu/CaregiverProjects